CLINICAL TRIAL: NCT04116502
Title: A Phase III, Randomised, Open-label, Multicenter International Trial Comparing Ruxolitinib With Either HydRoxycarbamIDe or Interferon Alpha as First Line ThErapy for High Risk Polycythemia Vera
Brief Title: MITHRIDATE: Ruxolitinib Versus Hydroxycarbamide or Interferon as First Line Therapy in High Risk Polycythemia Vera
Acronym: MITHRIDATE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Novartis (Industry); MPN Voice (Unknown); French National Cancer Institute (Institut National Du Cancer - France) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_16-148
Record Dates: First submitted 2019-09-09; First posted 2019-10-04 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera | interventions — ruxolitinib; Hydroxyurea; Interferon-alpha; Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A- Ruxolitinib (Experimental): Treatment with Ruxolitinib
  Interventions: Drug: Ruxolitinib
- B- Hydroxycarbamide OR Interferon A (Active Comparator): Best Available Therapy (BAT), Treatment with hydroxycarbamide OR Interferon A
  Interventions: Drug: Hydroxycarbamide; Drug: Interferon-Alpha

INTERVENTIONS:
Drug: Ruxolitinib — 10mg of ruxolitinib twice daily (bd)
  Other Names: Jakavi®
  Arms: A- Ruxolitinib
Drug: Hydroxycarbamide — Via standard hospital mechanisms
  Other Names: Hydroxyurea
  Arms: B- Hydroxycarbamide OR Interferon A
Drug: Interferon-Alpha — Any formulation, via standard hospital mechanisms
  Other Names: Interferon, alpha interferon, Intron® A, Roferon® A
  Arms: B- Hydroxycarbamide OR Interferon A

SUMMARY:
The trial will be a phase III, randomised-controlled, multi-centre, international, open-label trial consisting of ruxolitinib versus best available therapy, where best available therapy is a choice of interferon alpha, any formulation permitted (IFN) or hydroxycarbamide (HC), and which will be elected by the Investigator prior to randomisation.

DETAILED DESCRIPTION:
The trial will be a phase III, randomised-controlled, multi-centre, international, open-label trial consisting of ruxolitinib versus best available therapy, where best available therapy is a choice of interferon alpha, any formulation permitted (IFN) or hydroxycarbamide (HC), and which will be elected by the Investigator prior to randomisation.

There will be no cross-over either between arm A and B or between therapies on Arm B

HC and IFN will be provided as best available therapy, IFN can include standard of pegylated-interferon at Investigators discretion.

ELIGIBILITY:
Population:

High risk PV defined as WBC >11 x 10^9/l* AND at least ONE of the following

* Age >60 years
* Prior thrombosis or haemorrhage
* Platelet count >1000 x 10^9/l*
* Hypertension or diabetes requiring pharmacological therapy (*At any time since diagnosis)

Inclusion Criteria:

1. Patient ≥18 years of age
2. Diagnosis of PV meeting the WHO criteria within the past 15 years
3. Meets criteria of high risk* PV (see above for specific population)
4. Patients must have a screening haemoglobin of >8g/dl
5. Patients may have received antiplatelet agents and venesection
6. Patients may have received ONE cytoreductive therapy for PV less than 10 years (BUT they should not be resistant or intolerant to that therapy)
7. Able to provide written informed consent

Exclusion Criteria:

1. Diagnosis of PV > 15 years previously
2. Absence of JAK-2 mutation
3. Patients with any contraindications to any of the investigational medical products
4. Treatment with >1 cytoreductive therapy OR a cytoreductive treatment duration exceeding 10 years OR resistance/intolerance to that therapy
5. Active infection including Human Immunodeficiency Virus (HIV), hepatitis B, hepatitis C, autoimmune hepatitis, Tuberculosis
6. Pregnant or lactating patients (Women of childbearing potential must have a negative urine or blood Human Chorionic Gonadotropin pregnancy test prior to trial entry)
7. Patients with lactose allergies, hypersensitivities, or rare hereditary problems, of galactose intolerance, total lactase deficiency or glucose- galactose malabsorption
8. Patients with uncontrolled neuropsychiatric disorders
9. Patients with uncontrolled cutaneous cancers
10. Patients and partners not prepared to adopt highly effective contraception measures (if sexually active) whilst on treatment and for at least 6 months after completion of study medication
11. ECOG Performance Status Score ≥ 3
12. Uncontrolled rapid or paroxysmal atrial fibrillation, uncontrolled or unstable angina, recent (within the last 6 months) myocardial infarction or acute coronary syndrome or any clinically significant cardiac disease > NYHA ( New York Heart Association) Class II
13. Patients who have transformed to myelofibrosis
14. Previous treatment with ruxolitinib
15. Previous (within the last 12 months) or current platelet count <100 x 109/L or neutrophil count < 1 x 109/L not due to therapy
16. Inadequate liver function as defined by ALT/AST >2.0 x ULN
17. Inadequate renal function as defined by eGFR < 30 mls/min
18. Unable to give informed consent

    Additional Exclusion Criteria for France Only
19. All women of childbearing potential (as per Appendix 8 definition)
20. No affiliation with the French healthcare system
21. Persons under psychiatric care that would impede understanding of informed consent and optimal treatment and follow-up
22. Adults subject to a legal protection measure (guardianship, curatorship and safeguard of justice)
23. Patients deprived of their liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | the time from randomisation to the date of the first major thrombosis/haemorrhage, death,transformation to Myelodysplastic Syndromes, Acute Myeloid Leukaemia or Post-polycythemia Vera Myelofibrosis, if within the ~3 year trial period
  Event Free Survival

SECONDARY OUTCOMES:
Major thrombosis | Occurring while on treatment (over 3 years)
  As defined in the protocol, combined and split to venous and arterial
Major haemorrhage | Occurring while on treatment (over 3 years)
  As defined in the protocol
Transformation to PPV-MF | Occurring while on treatment (over 3 years)
  Transformation to PPV-MF
Transformation to MDS and/or AML | Occurring while on treatment (over 3 years)
  Transformation to MDS and/or AML
Complete Haematological remission (CHR) | 1 year post-treatment
  As defined by ELN response criteria at 1 year
Symptom burden/Quality of life (MPN-SAF) | Questionnaires collected at baseline, weeks 12, 26, 39, 55, months 15, 18, 24, 30 and 36
  As measured via MPN-SAF
Symptom burden/Quality of life (MDASI) | Questionnaires collected at baseline, weeks 12, 26, 39, 55, months 15, 18, 24, 30 and 36
  As measured via MDASI
Symptom burden/Quality of life (EQ-5D) | Questionnaires collected at baseline, weeks 12, 26, 39, 55, months 15, 18, 24, 30 and 36
  As measured via EQ-5D
Health economics | At the end of the trial (trial duration of approximately 8 years)
  Including cost utility and cost effectiveness analyses as defined by the protocol (e.g. QALYs)
Peripheral blood JAK2 V617F allele burden | At baseline and annually throughout the trial (from baseline until approximately 3 years post-randomisation)
  According to ELN response criteria
Rates of discontinuation | From treatment prior to protocol defined 3 years
  Trial discontinuation
Rate and severity of adverse events | Continuous throughout the trial (from randomisation until approximately 3 years post-randomisation))
  collected according to CTCAE version 4.0 and the MITHRIDATE protocol
Spleen response | Response at 1 year post randomisation
  in patients with splenomegaly
Time free from venesection | Defined as the mean time between venesections while on trial treatment (treatment duration of 3 years)
  Time free from venesection
Secondary malignancy | Occurring throughout the trial (from randomisation until approximately 3 years post-randomisation)
  Malignancy independent to the original diagnosis
Change in QRisk score | Collected at baseline and years 1, 2 and 3
  Change in QRisk score

OTHER OUTCOMES:
Progression of marrow fibrosis | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  Progression of marrow fibrosis (bone marrow collected and analysed at the Weatherall Institute of Molecular Medicine (WIMM) in Oxford
Impact of treatment on molecular signatures of disease | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  Impact of treatment on molecular signatures of disease (as analysed by the WIMM in Oxford)
Clonal involvement | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  within the stem/progenitor cell compartment (as analysed by the WIMM in Oxford)
Clonal evolution | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  (acquisition of additional mutations, as analysed by the WIMM in Oxford)
Reduction of peripheral blood allele burden | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  of other disease-association mutations (as analysed by the WIMM in Oxford)
Assessment of the prevalence of clonality markers for haematological disease | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  and any change over time (as analysed by the WIMM in Oxford)
Cardiac event | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  (angina, acute coronary syndrome, acute MI; arrhythmia)
Pulmonary hypertension | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  Pulmonary hypertension as assessed clinically
Coronary intervention | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  e.g. angiogram, angioplasty, CABG
Deterioration in cardiac function | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  e.g. LVEF% on ECHO/MUGA and/or NYHA classification
Cerebrovascular event | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  TIA, haemorrhagic CVA, non-haemorrhagic CVA
Arterial vascular event | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  peripheral vascular disease: claudication, carotid stenosis
Venous thrombosis | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  including DVT, PE, Cerebral, splanchnic, other
Pregnancy loss | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  Pregnancy loss
Thrombosis biomarkers | Occurring throughout the trial (from randomisation to approximately 3 years post-randomisation)
  Correlation of thrombosis biomarkers with clinical thrombosis events

CONTACTS AND LOCATIONS:
Overall Officials: Claire Harrison, Principal Investigator — Acting on behalf of the Sponsor (UK), Guy's Hospital, London, UK, SE1 9RT; Jean-Jacques Kiladjian, Principal Investigator — (France) Clinical Investigations Center, Saint-Louis Hospital, Paris, France
Locations (47):
- United Kingdom (47):
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal United Hospital, Bath
  - Belfast City Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - Royal Bournemouth Hospital, Bournemouth
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - University Hospital of Wales, Cardiff
  - St Richard's Hospital, Chichester
  - Colchester Hospital, Colchester
  - Castle Hill Hospital, Cottingham
  - Russells Hall Hospital, Dudley
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Gloucestershire Royal Hospital, Gloucester
  - Calderdale Royal Hospital, Halifax
  - Huddersfield Royal Infirmary, Huddersfield
  - Raigmore Hospital, Inverness
  - Kettering General Hospital, Kettering
  - Leicester Royal Infirmary, Leicester
  - St John's Hospital, Livingston
  - University College Hospital, London
  - Guy's Hospital, London
  - St George's Hospital, London
  - Wythenshawe Hospital, Manchester
  - Arrowe Park Hospital, Metropolitan Borough of Wirral
  - The James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Royal Gwent Hospital, Newport
  - North Tyneside General Hospital, North Shields
  - Northampton General Hospital, Northampton
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Royal Berkshire Hospital, Reading
  - Halton Hospital, Runcorn
  - Wexham Park Hospital, Slough
  - Southampton General Hospital, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Sunderland Royal Hospital, Sunderland
  - Good Hope Hospital, Sutton Coldfield
  - Royal Cornwall Hospital, Truro
  - Warwick Hospital, Warwick
  - New Cross Hospital, Wolverhampton
  - Worthing Hospital, Worthing

IPD SHARING:
Plan to Share IPD: No